CLINICAL TRIAL: NCT00398372
Title: Le20: Clinical and Pathologic Studies in Non-Hodgkin's Lymphoma Patients Receiving Antibody Treatment
Brief Title: Clinical and Pathologic Studies in Non-Hodgkin's Lymphoma Patients Receiving Antibody Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Amgen (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Wen-Kai Weng, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: LYMNHL0031; 200114861; 77550; CA09287; CA111827; LYMNHL0031; NCT00398372
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2010-07

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphomas: Non-Hodgkin; Lymphomas: Non-Hodgkin Cutaneous Lymphoma; Lymphomas: Non-Hodgkin Diffuse Large B-Cell; Lymphomas: Non-Hodgkin Follicular / Indolent B-Cell; Lymphomas: Non-Hodgkin Mantle Cell; Lymphomas: Non-Hodgkin Marginal Zone; Lymphomas: Non-Hodgkin Peripheral T-Cell; Lymphomas: Non-Hodgkin Waldenstr Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; epratuzumab

INTERVENTIONS:
Drug: Rituximab
Drug: Epratuzumab

SUMMARY:
To characterize the molecular and cell biology of the tumor cells in lymphoma. The mechanism of monoclonal antibody treatment by rituximab or epratuzumab will also be examined.

ELIGIBILITY:
Inclusion Criteria:Non-Hodgkin's Lymphoma Patients Receiving Antibody Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2000-11; Primary Completion 2007-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To characterize the molecular and cell biology of the tumor cells in lymphoma. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kai Weng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States